CLINICAL TRIAL: NCT07247305
Title: Screen Culture's Impact on Generation Z Adolescents' Physical Activity, Posture and Well-being in Egypt: A Cross-sectional Study
Brief Title: Screen Culture's Impact on Generation Z Adolescents' Physical Activity, Posture and Well-being in Egypt
Status: Not yet recruiting | Type: Observational
Sponsor: Sinai University (Other)
Responsible Party: Principal Investigator, Alaa Noureldeen Kora, Lecturer , Principal Investigator, Sinai University
Other Study IDs: SU.REC.2024 (57 H)
Record Dates: First submitted 2025-11-14; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Adolescence; Adolescent; Well Being; Posture; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolesence: Age: 13-18 years (adolescence as per WHO standards).
  * Nationality: Egyptian residents.
  * Language Proficiency: Ability to read and comprehend English (the questionnaires are in English).
  Interventions: Diagnostic Test: BMI Measurement; Diagnostic Test: Screen Time Questionnaire (QUEST); Diagnostic Test: Insomnia Severity Index (ISI); Diagnostic Test: Q-BAPHYP; Diagnostic Test: PedsQL™

INTERVENTIONS:
Diagnostic Test: BMI Measurement — BMI Measurement: Self-report height/weight (compared with age/sex standard BMI percentiles).
Diagnostic Test: Screen Time Questionnaire (QUEST) — Screen Time Questionnaire (QUEST): Assess length, purpose, and pattern of device use.
Diagnostic Test: Insomnia Severity Index (ISI) — Insomnia Severity Index (ISI): 7-item sleep disturbance severity measure (score range: 0-28).
Diagnostic Test: Q-BAPHYP — Q-BAPHYP: 20-item scale measuring body awareness, postural habits, and ergonomic behaviors.
Diagnostic Test: PedsQL™ — PedsQL™: Pediatric Quality of Life Inventory

SUMMARY:
Ubiquitous adoption of screen-based technologies has transformed the behavioral and physiological environment of Generation Z youth. In Egypt, where digital adoption speeds up with apace urbanisation, teens (13-18) have greater exposure to computers, mobile phones, and other screen-based devices.

Growing evidence points towards excessive viewing of screens in compromised well-being, including sleep issues, inactive lifestyles, weight loss/gain, and musculoskeletal disturbances. Contextual evidence for the Egyptian teenager is scarce.

This study fills the gap by investigating the multi-dimensional influence of screen culture on physical well-being, focusing on sleep quality, body mass index (BMI), posture, physical activity, and disability outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age: 13-18 years (adolescence as per WHO standards).
* Nationality: Egyptian residents.
* Language Proficiency: Ability to read and comprehend English (the questionnaires are in English).
* Screen Use: ≥1 screen device used frequently (e.g., smartphone, laptop, tablet).

Exclusion Criteria:

* Can not o read and comprehend English language Do not have a routine of a screen time

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Generation Z Adolescences (Age 13 to 18)
Sampling Method: Probability Sample
Enrollment: 385 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
sleep disturbance severity | 1 day
  Scale Used: Insomnia Severity Index (ISI)
  Description:
  The ISI is a 7-item self-report questionnaire that assesses the severity of insomnia and its impact on daily functioning. Each item is scored on a 0-4 scale, with total scores ranging from 0 to 28. Higher scores indicate more severe sleep disturbance.
body awareness | 1 Day
  Scale Used: Q-BAPHYP
  Description:
  The body awareness component of the Q-BAPHYP scale assesses an individual's awareness of their body position, movement, and physical sensations. It may include items related to:
  Recognition of poor posture
  Awareness of physical discomfort during screen use
  Sensitivity to bodily signals (e.g., fatigue, muscle tension)
  Attention to ergonomic positioning
Pediatric Quality of Life | 1 Day
  Scale Used: PedsQL™ (Pediatric Quality of Life Inventory)
  Description:
  The PedsQL™ is a modular instrument designed to measure health-related quality of life in children and adolescents. It covers multiple dimensions of well-being across:
  Physical Functioning (e.g., ability to engage in physical activities)
  Emotional Functioning (e.g., feeling anxious or sad)
  Social Functioning (e.g., interactions with peers)
  School Functioning (e.g., ability to concentrate and attend school)

SECONDARY OUTCOMES:
Postural Habits | 1 Day
  The body awareness component of the Q-BAPHYP scale assesses an individual's awareness of their body position, movement, and physical sensations

CONTACTS AND LOCATIONS:
Locations (1):
- Sinai University, Ismailia, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
According to the data confidentiality

REFERENCES:
- [Result] Priftis N, Panagiotakos D. Screen Time and Its Health Consequences in Children and Adolescents. Children (Basel). 2023 Oct 8;10(10):1665. doi: 10.3390/children10101665. PMID 37892328
- [Result] Fan H, Yan J, Yang Z, Liang K, Chen S. Cross-sectional associations between screen time and the selected lifestyle behaviors in adolescents. Front Public Health. 2022 Sep 27;10:932017. doi: 10.3389/fpubh.2022.932017. eCollection 2022. PMID 36238246
- [Result] Badran M. Young people and the digital divide in Egypt: an empirical study. Eurasian Econ Rev. 2014;4:223-50.
- [Result] Armaneous A, Atta H, ElKhatib A, Kamal A, Sallam S. Internet Addiction among Egyptian Teens during COVID-19 Pandemic. Open Access Maced J Med Sci. 2024;12:388-97.
- [Result] Stiglic N, Viner RM. Effects of screentime on the health and well-being of children and adolescents: a systematic review of reviews. BMJ Open. 2019 Jan 3;9(1):e023191. doi: 10.1136/bmjopen-2018-023191. PMID 30606703